CLINICAL TRIAL: NCT01282957
Title: Financial Incentives for Home-based Health Management: A Pilot Randomized Trial
Brief Title: Way to Health, Healthy Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 812211; RC2AG036592 (NIH)
Record Dates: First submitted 2011-01-10; First posted 2011-01-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Control (No Intervention): Daily use of three home-monitoring devices: glucometer, blood pressure cuff and scale for 6 months
- Financial Incentive Group I (Experimental): Daily use of three home-monitoring devices: glucometer, blood pressure cuff and scale for 3 months. If all three devices used daily, participant entered in lottery with 1 in 100 odds of winning $100 and 2 in 10 odds of winning $10. Financial incentive terminated after 3 months. Daily use of devices continues for additional 3 months. (Intervention involves the daily lottery itself along with feedback via email or text messaging to participants about the lottery results and whether or not they were included based on device adherence.)
  Interventions: Behavioral: Financial Incentive Group I
- Financial Incentives Group II (Experimental): Daily use of three home-monitoring devices: glucometer, blood pressure cuff and scale for 3 months. If all three devices used daily, participant entered in lottery with 1 in 100 odds of winning $50 and 2 in 10 odds of winning $5. Financial incentive terminated after 3 months. Daily use of devices continues for additional 3 months. (Intervention involves the daily lottery itself along with feedback via email or text messaging to participants about the lottery results and whether or not they were included based on device adherence.)
  Interventions: Behavioral: Financial Incentive Group II

INTERVENTIONS:
Behavioral: Financial Incentive Group I — Lottery with 1 in 100 odds of $100 and 18 in 100 odds of $10. The intervention involves the daily lottery itself along with feedback via email or text messaging to participants about the lottery results and whether or not they were included based on device adherence.
  Arms: Financial Incentive Group I
Behavioral: Financial Incentive Group II — Lottery with 1 in 100 odds of $50 and 18 in 100 odds of $5. The intervention involves the daily lottery itself along with feedback via email or text messaging to participants about the lottery results and whether or not they were included based on device adherence.
  Arms: Financial Incentives Group II

SUMMARY:
The primary objective of the study is to assess the effect of financial incentives on the use of home health monitoring devices among high-risk patients. In addition, there are three secondary objectives: (1) obtain preliminary evidence regarding whether the monetary value of incentives has a differential effect on the use of home health monitoring devices; (2) identify potential barriers that prohibit regular use of home-based health devices using qualitative data; and (3) assess the usability of a newly developed web portal and its feasibility for future randomized clinical trials aimed at changing health-related behaviors.

DETAILED DESCRIPTION:
While home monitoring of health appears to be a promising frontier in health care, patient adherence to, and utilization of, such devices is often low, limiting the potential benefit of this technology. Financial incentives have been effective in increasing rates of weight loss, smoking cessation, and medication adherence and therefore may increase rates of utilization of home-based health monitoring devices. Therefore, in this study, we test the effects of lottery-based incentives on use of home-based health monitoring technologies.

The aim of this pilot randomized controlled trial is to evaluate whether financial incentives delivered through a novel online platform can effectively increase use of home-based health monitoring technology among overweight adults with diabetes. Our primary objective is to assess the effects of financial incentives on the use of home health monitoring devices among high-risk patients. In addition, we have three secondary objectives: (1) obtain preliminary evidence regarding whether the monetary value of incentives has a differential effect on the use of home health monitoring devices; (2) identify potential barriers that prohibit regular use of home-based health devices using qualitative data; and (3) assess the usability of a newly developed web portal and its feasibility for future randomized clinical trials aimed at changing health-related behaviors.

Participants will be randomized into each of the following three arms: (1) Financial Incentive Group I; (2) Financial Incentive Group II; (3) Control Group. Incentives for Financial Groups I and II are designed in a way that builds on the success of previous incentive-based interventions for weight loss. Both lotteries are tailored to provide infrequent large payoffs and frequent small payoffs since lottery players are motivated by both the possibility of a large reward and the opportunity for regular, immediate rewards. The average expected payoff value of Financial Incentive Group I will be $2.80 per day and $1.40 per day in Financial Incentive Group II. The interventions will run for 91 days starting at randomization. At the end of the intervention time period, each participant will be notified that the intervention period has ended and the 90-day follow-up period has begun. During the follow-up period each participant will continue to upload measurements daily, but will not receive incentives or reminders.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 80 years of age
* Hemoglobin A1c measured in the last six weeks greater than or equal to 7.5%
* Weight less than 425lbs
* Cell phone with text messaging capabilities or email access
* Followed by Primary Care Provider at Penn Internal Medicine Associates practice at 3701 Market St

Exclusion Criteria:

* Lack or are unwilling to use email or cell phone for text messaging
* Are enrolled in other, ongoing clinical trials
* Suffer from an uncontrolled psychiatric disease
* Have a history or diagnosis of heart failure as confirmed by ICD-9 codes: 428.0 (congestive heart failure), 425.0 (cardiomyopathy), and 414.8 ischemic cardiomyopathy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Rate of use of the three home-based technologies | 3-months
  We will analyze the proportion of days that home monitoring was completed (defined as successful reporting of data from all three devices - weight, blood pressure and blood sugar) compared to failure to report across all groups after the end of the 3-month intervention period.

SECONDARY OUTCOMES:
Usability and functionality of the study's online web portal, Way to Health, and wifi-enabled home health monitoring devices | 6-months
  We will ask participants to participate in a qualitative interview at the final study visit to assess the usability and functionality of the web portal and study devices for use during future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Derived] Sen AP, Sewell TB, Riley EB, Stearman B, Bellamy SL, Hu MF, Tao Y, Zhu J, Park JD, Loewenstein G, Asch DA, Volpp KG. Financial incentives for home-based health monitoring: a randomized controlled trial. J Gen Intern Med. 2014 May;29(5):770-7. doi: 10.1007/s11606-014-2778-0. Epub 2014 Feb 13. PMID 24522623